CLINICAL TRIAL: NCT00147134
Title: Randomized Controlled Trial to Evaluate Laparoscopic Versus Open Surgery for Colorectal Cancer（JCOG 0404,CRC Surg-LAP/OPEN)
Brief Title: A Trial to Evaluate Laparoscopic Versus Open Surgery for Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0404; C000000105
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; laparoscopic surgery; randomized controlled trial; oncological outcome
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Procedure/Surgery: open colectomy
  Interventions: Procedure: open colectomy
- 2 (Experimental): Procedure/Surgery: laparoscopic colectomy
  Interventions: Procedure: laparoscopic colectomy

INTERVENTIONS:
Procedure: open colectomy — Procedure/Surgery: open colectomy
  Arms: 1
Procedure: laparoscopic colectomy — Procedure/Surgery: laparoscopic colectomy
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate oncological outcome of patients for T3 and T4 colorectal cancer undergoing laparoscopic versus open surgery.

DETAILED DESCRIPTION:
The benefits of laparoscopic surgery (LAP) in comparison to open surgery (OPEN) have been suggested with respect to decreased morbidity, decreased pain, faster recovery, and shorter hospital stay.1-4 However, the long-term survival of LAP for colorectal cancer is still unclear, especially for advanced colorectal cancer requiring extended lymphadenectomy. Thus, the investigators designed a study which investigates whether LAP is suitable for advanced colorectal cancer with respect to survival and post-operative morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven colorectal carcinoma
2. Tumor located in the cecum, ascending colon, sigmoid colon, or rectosigmoid colon
3. T3 or deeper lesion without involvement of other organs
4. Without multiple lesion other than carcinoma in situ
5. Cancer classified as N0-2 and M0, according to the TNM classification system
6. Tumor size < 8 cm
7. No bowel obstruction
8. Age 20 < and > 75 years
9. Sufficient organ function
10. No history of gastrointestinal surgery
11. No history of chemotherapy or radiotherapy
12. Provided written informed consent

Exclusion Criteria:

1. Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ
2. Severe pulmonary emphysema, interstitial pneumonitis, or ischemic heart disease
3. Pregnant or lactating women
4. Severe mental disease
5. Continuous systemic steroid therapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2004-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | During the study conduct

SECONDARY OUTCOMES:
Relapse-free survival | During the study conduct
Short-term clinical outcomes | time to 1st discharge after operation
Adverse events | During the study conduct
The proportion of conversion from LAP to OPEN | operation day
The proportion of completion of LAP | operation day

CONTACTS AND LOCATIONS:
Overall Officials: Seigo Kitano, MD, PhD,FACS, Study Chair — Oita University
Locations (26):
- Japan (26):
  - Fujita Health University, Toyoake,Kutsukake-cho,Dengakugakubo,1-98, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - Toho University Sakura Hospital, Sakura,Shimoshidu,564-1, Chiba
  - Jyuntendo Urayasu Hospital, Urayasu,Tomioka,2-1-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kurume University School of Medicine, Kurume,Asahi-machi,67, Fukuoka
  - Hiroshima University, School of Medicine, Hiroshima,Minami-ku,Kasumi,1-2-3, Hiroshima
  - Ishikawa Prefectual Central Hospital, Kanazawa,Kuratsuki-Higashi,2-1, Ishikawa-ken
  - Teikyo University Hospital, Mizonokuchi, Kawasaki,Takatsu-ku,Mizonokuchi,3-8-3, Kanagawa
  - Kitasato University East Hospital, Sagamihara,Asamizodai,2-1-1, Kanagawa
  - Kitasato University School of Medichine, Sagamihara,Kitasato,1-15-1, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama,Tsuzuki-ku,Chigasakichuo,35-1, Kanagawa
  - National Hospital Organization Kyoto Medical Center, Kyoto,Fushimi-ku,Fukakusa,Mukaihata-cho,1-1, Kyoto
  - Nagano Municipal Hospital, Nagano,Tomitake,1333-1, Nagano
  - Oita University Faculty of Medicine, Yufu city,Hasama-machi, 1-1, Oita Prefecture
  - Osaka City General Hospital, Osaka,Miyakojima-ku,Miyakojimahondori,2-13-22, Osaka
  - Osaka University Graduate School of Medicine, Suita,Yamada-oka,2-2, Osaka
  - Osaka Medical College, Takatsuki,Daigakucho,2-7, Osaka
  - Omiya Medical Center, Jichi Medical School, Saitama,Omiya-ku,Amanuma-cho,1-847, Saitama
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku,Yushima,1-5-45, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Toho University Ohashi Hospital, Meguro-ku,Ohashi,2-17-6, Tokyo
  - Toranomon Hospital, Minato-ku,Toranomon,2-2-2, Tokyo
  - Kyorin University School of Medicine, Mitaka,Shinkawa,6-20-2, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo

REFERENCES:
- [Derived] Saito S, Akagi T, Katayama H, Wakabayashi M, Inomata M, Yamamoto S, Ito M, Kinugasa Y, Egi H, Munakata Y, Kokuba Y, Bando H, Yasui M, Ikeda M, Nakajima K, Shida D, Kanemitsu Y, Kitano S; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Identification of patient subgroups with unfavorable long-term outcomes associated with laparoscopic surgery in a randomized controlled trial comparing open and laparoscopic surgery for colon cancer (Japan Clinical Oncology Group Study JCOG0404). Ann Gastroenterol Surg. 2021 Aug 9;5(6):804-812. doi: 10.1002/ags3.12475. eCollection 2021 Nov. PMID 34755012
- [Derived] Nishizawa Y, Akagi T, Inomata M, Katayama H, Mizusawa J, Yamamoto S, Ito M, Masaki T, Watanabe M, Shimada Y, Kitano S. Risk factors for early postoperative complications after D3 dissection for stage II or III colon cancer: Supplementary analysis of a multicenter randomized controlled trial in Japan (JCOG0404). Ann Gastroenterol Surg. 2019 Apr 4;3(3):310-317. doi: 10.1002/ags3.12246. eCollection 2019 May. PMID 31131360
- [Derived] Fujii S, Akagi T, Inomata M, Katayama H, Mizusawa J, Ota M, Saito S, Kinugasa Y, Yamaguchi S, Sato T, Kitano S; Japan Clinical Oncology Group. Transitional impact of short- and long-term outcomes of a randomized controlled trial to evaluate laparoscopic versus open surgery for colorectal cancer from Japan Clinical Oncology Group Study JCOG0404. Ann Gastroenterol Surg. 2019 Mar 26;3(3):301-309. doi: 10.1002/ags3.12245. eCollection 2019 May. PMID 31131359
- [Derived] Kitano S, Inomata M, Mizusawa J, Katayama H, Watanabe M, Yamamoto S, Ito M, Saito S, Fujii S, Konishi F, Saida Y, Hasegawa H, Akagi T, Sugihara K, Yamaguchi T, Masaki T, Fukunaga Y, Murata K, Okajima M, Moriya Y, Shimada Y. Survival outcomes following laparoscopic versus open D3 dissection for stage II or III colon cancer (JCOG0404): a phase 3, randomised controlled trial. Lancet Gastroenterol Hepatol. 2017 Apr;2(4):261-268. doi: 10.1016/S2468-1253(16)30207-2. Epub 2017 Feb 2. PMID 28404155
- [Derived] Yamamoto S, Inomata M, Katayama H, Mizusawa J, Etoh T, Konishi F, Sugihara K, Watanabe M, Moriya Y, Kitano S; Japan Clinical Oncology Group Colorectal Cancer Study Group. Short-term surgical outcomes from a randomized controlled trial to evaluate laparoscopic and open D3 dissection for stage II/III colon cancer: Japan Clinical Oncology Group Study JCOG 0404. Ann Surg. 2014 Jul;260(1):23-30. doi: 10.1097/SLA.0000000000000499. PMID 24509190
- See also: Related Info — http://www.jcog.jp/